CLINICAL TRIAL: NCT00245232
Title: Cognitive Processes in PTSD: Treatment
Brief Title: Cognitive Processing Therapy Versus Its Individual Components in the Treatment of Post-Traumatic Stress Disorder and Depression in Women Who Have Been Sexually Abused
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Missouri, St. Louis (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: R01MH051509-06 (NIH); R01MH051509-06 (NIH); DSIR AT-AS
Record Dates: First submitted 2005-10-25; First posted 2005-10-27 (Estimated); Last update posted 2015-03-31 (Estimated); Status verified 2015-03

CONDITIONS: Post-Traumatic Stress Disorder
Keywords: PTSD; Cognitive therapy; Rape
MeSH Terms: conditions — Stress Disorders, Post-Traumatic | interventions — Cognitive Behavioral Therapy

INTERVENTIONS:
Behavioral: Cognitive Therapy
Behavioral: Cognitive Processing Therapy
Behavioral: Written Exposure

SUMMARY:
This study will evaluate the effectiveness of cognitive processing therapy versus its individual components in treating women with post-traumatic stress disorder (PTSD) and depression brought on by sexual assault.

DETAILED DESCRIPTION:
PTSD is a psychiatric disorder that can occur following exposure to a traumatic event in which grave physical harm occurred or was threatened. PTSD is marked by clear biological changes as well as psychological symptoms. Many people with PTSD repeatedly relive the trauma in the form of flashback episodes, memories, nightmares, or frightening thoughts. This study will evaluate the effectiveness of cognitive processing therapy versus its individual components in treating women with post-traumatic stress disorder and depression brought on by sexual assault.

Participants in this single-blind study will be randomly assigned to receive one of three treatments: cognitive processing therapy (CPT); cognitive therapy (CT); or written exposure (WE). Participants assigned to receive either CPT or CT will attend therapy sessions twice weekly for 6 weeks. CPT will focus on helping each individual to process accurate memories of the traumatic event and to work through any memories that cannot be completely ignored, nor completely integrated back into their thinking. Also included in CPT will be a WE component, in which participants will be encouraged to recall the traumatic event and experience any emotions connected to it. CT will be similar to CPT, but will not include the WE component. Participants assigned to receive only WE will attend one 2-hour session each week. Symptoms of PTSD and depression will be measured at baseline, post-treatment, and at a 6-month follow-up visit.

ELIGIBILITY:
Inclusion Criteria:

* History of a discrete episode of assault in childhood or adulthood
* Meets criteria for post-traumatic stress disorder

Exclusion Criteria:

* Experienced a traumatic event that was in the form of chronic ongoing abuse and not a discrete incidence
* Psychosis
* Mental retardation
* Suicidal or parasuicidal
* Currently addicted to drugs
* Illiterate
* Currently in an abusive relationship
* Currently being stalked

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 228
Dates: Start 2000-08; Study Completion 2005-04

PRIMARY OUTCOMES:
Depression symptoms; measured immediately post-treatment and 6 months post-treatment
Post-traumatic stress disorder symptoms; measured immediately post-treatment and 6 months post-treatment

CONTACTS AND LOCATIONS:
Overall Officials: Patricia A. Resick, PhD, Principal Investigator — National Center for PTSD, Women's Health Sciences Division
Locations (1):
- Center for Trauma and Recovery, University of Missouri - St. Louis, St Louis, Missouri, United States

REFERENCES:
- [Result] Resick PA, Nishith P, Weaver TL, Astin MC, Feuer CA. A comparison of cognitive-processing therapy with prolonged exposure and a waiting condition for the treatment of chronic posttraumatic stress disorder in female rape victims. J Consult Clin Psychol. 2002 Aug;70(4):867-79. doi: 10.1037//0022-006x.70.4.867. PMID 12182270
- [Derived] O'Doherty L, Whelan M, Carter GJ, Brown K, Tarzia L, Hegarty K, Feder G, Brown SJ. Psychosocial interventions for survivors of rape and sexual assault experienced during adulthood. Cochrane Database Syst Rev. 2023 Oct 5;10(10):CD013456. doi: 10.1002/14651858.CD013456.pub2. PMID 37795783
- [Derived] Fitzpatrick SS, Liebman RE, Monson CM, Resick PA. Latent emotion profiles of PTSD and specific emotions predicting differential therapy outcomes in a dismantling study of cognitive processing therapy. J Anxiety Disord. 2023 Apr;95:102681. doi: 10.1016/j.janxdis.2023.102681. Epub 2023 Feb 17. PMID 36848714